CLINICAL TRIAL: NCT05461027
Title: Percutaneous Cryoablation of Central Kidney Tumours With Temporary Renal Artery Occlusion
Acronym: CP-Renal
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8529
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Kidney Cancer
Keywords: Kidney Cancer; Central Kidney Tumours; Renal Artery Occlusion; cryoablation; Urological surgery; T1a tumours; Cold sink effect; Endovascular balloon clamping; Renal hilum
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Percutaneous cryoablation is an alternative to urological surgery for T1a tumours, whose oncological efficacy decreases for the most central tumours due to a cold sink effect.

ELIGIBILITY:
Inclusion criteria:

* Adult subject (≥18 years)
* Subject who has undergone cryoablation of a central kidney tumour with temporary occlusion of the renal artery by an endovascular balloon at the HUS during the period 01/01/2018 to 30/12/2021
* Subject who has not expressed his/her opposition, after information, to the re-use of his/her data for the purpose of this research.

Exclusion criteria :

* Subject having expressed his/her opposition to participate in the study
* Subject under legal protection, guardianship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult subject (≥18 years) who has undergone cryoablation of a central kidney tumour with temporary occlusion of the renal artery by an endovascular balloon at the HUS during the period 01/01/2018 to 30/12/2021
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Description of the technique of percutaneous cryoablation of central renal tumours with temporary balloon obliteration of the renal artery | Files analysed retrospectively from January 01, 2018 to December 31, 2021 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Alexis AUTRUSSEAU, MD, Principal Investigator — Service d'Imagerie Interventionnelle - CHU de Strasbourg - France
Locations (1):
- Service d'Imagerie Interventionnelle - CHU de Strasbourg - France, Strasbourg, France